CLINICAL TRIAL: NCT03228563
Title: The Effect of Probiotics on Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, I-Kuan Wang, Attending physician, China Medical University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH106-REC1-015
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Chronic Kidney Disease; Probiotics; Renal Function
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Taking two capsules of probiotics twice daily for 12 months.
  Interventions: Other: Probioics
- Healthy control (No Intervention): Healthy volunteers were: no hypertension (Blood pressure<140/90mmHg), no diabetes (Glucose AC 70~100mg/dl), no hyperlipidemia (Cholesterol Total 130~200mg/dL、Triglyceride<150mg/dL), no urinary protein (-) and normal renal function (eGFR>90), after signing the consent form, the stool samples will be collected.

INTERVENTIONS:
Other: Probioics — CKD Patients were supplemented with two capsules of probiotics containing 2.5*10^9 CFU Lactobacillus acidophilus (TYCA06), Bifidobacterium longum (BLI-02) and Bifidobacterium bifidum (VDD088) twice daily for 12 months.
  Arms: Probiotics

SUMMARY:
Probiotics could attenuate renal function deterioration in CKD patients.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a global health issue that has a substantial impact on affected individuals. Chronic inflammation, which is widely seen in CKD including long-term dialysis patients, is associated with malnutrition, atherosclerosis and an increased mortality risk. Inflammatory markers such as C-reactive protein, IL-6, IL-18, and TNF-α, are elevated in dialysis patients and can predict cardiovascular event and all-cause mortality. Endotoxin is bacterial lipopolysaccharide, and makes up the outer membrane of Gram-negative bacteria. Endotoxin is also an important source and also a marker of inflammation in CKD.

The natural intestinal microbiota is altered in CKD patients as an increase in aerobic bacteria such as E. coli and a decrease in anaerobic bacteria such as Bifidobacterium. Dysbiosis might contribute to the chronic inflammatory state in dialysis patients through endotoxemia, induction of the pro-inflammatory cytokine, and production of uremic toxins through fermentation of protein in the large intestine. Probiotics containing Bifidobacterium species and Lactobacilli species could benefit the host by inhibiting the growth or epithelial invasion of pathogenic bacteria, enhancing the intestinal barrier function, and regulating the immune system.

Probiotics could suppress proinflammatory cytokines, such as TNF-α and IL-6 . In addition, probiotics could improve renal function parameters in uremic rats and significantly lower levels of blood urea nitrogen in stage 3 and 4 CKD patients. The aim of the present study is to evaluate:

1. Whether probiotics could retard the decline of renal function?
2. Whether probiotics could change microbiota?
3. Whether probiotics could reduce the serum levels of endotoxin and cytokines (TNF-α, IL-6, and IL-18)?
4. Whether probiotics could improve the gastrointestinal symptoms in CKD patients?

Estimated glomerular filtration rate, stool microbiota, serum cytokines and endotoxin, and gastrointestinal symptoms of stage 3-5 patients are measured before and after intervention. The Wilcoxon signed-rank and Wilcoxon rank-sum tests were used to compare intra- and intergroup differences for continuous variables, as appropriate. A p value less than 0.05 was considered significant.

ELIGIBILITY:
Healthy volunteers:

The criteria for healthy volunteers were: no hypertension (Blood pressure<140/90mmHg), no diabetes (Glucose AC 70~100mg/dl), no hyperlipidemia (Cholesterol Total 130~200mg/dL、Triglyceride<150mg/dL), no urinary protein (-) and normal renal function (eGFR>90), after signing the consent form, the stool samples will be collected.

CKD patients:

Inclusion Criteria:

‧Stage 3-5 CKD patients, at least 20 years of age and regular follow-up for at least 6 months prior to enrollment.

Exclusion Criteria:

* Pregnancy.
* On immunosuppressive therapy.
* Active infectious condition.
* Acute kidney injury.
* Consuming other forms of probiotics.
* Taking antibiotics within 30 days prior to enrollment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
eGFR decline rate. | 12 months.
  Compare estimated glomerular filtration rate decline rate within baseline, 3, 6, 9 and 12 months after taking probiotics.

SECONDARY OUTCOMES:
Change rate in serum pro-inflammatory cytokines (TNF-α, IL6 and IL18) and endotoxin. | 12 months
  Compare TNF-α, IL6, IL18 and endotoxin concentration within baseline, 3, 6, 9 and 12 months after taking probiotics.
Average scores of gastrointestinal symptoms by questionnaire. | 12 months.
  Gastrointestinal symptoms are evaluated by a study nurse using questionnaire at baseline, 3, 6, 9 and 12 months after intervention. The questionnaire included the stool form [1 = very hard (small hard lumps), 2 = hard stool (hard sausage shape), 3 = normal stool (sausage to banana shape), 4 = soft stool, 5 = muddy stool, 6 = watery stool], ease of defecation (1 = difficult, 2 = easy, 3 = very easy) and abdominal symptoms [frequency of upper abdominal pain, lower abdominal pain, borborygmus, and flatulence (1 = frequent, 2 = occasional, 3 = almost never)]. The average scores before and after the intervention were analyzed.
Relative abundance of intestinal microbiota. | 12 months.
  Stools from the participants were collected before and after 3, 6, 9 and 12-month probiotics treatments for NGS assay. The abundance of Bifidobacterium and Lactobacillus in stool microbiotia will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: I-kuan Wang, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan